CLINICAL TRIAL: NCT00492778
Title: A Randomized Trial of Pelvic Irradiation With or Without Concurrent Weekly Cisplatin in Patients With Pelvic-Only Recurrence of Carcinoma of the Uterine Corpus
Brief Title: Radiation Therapy With or Without Cisplatin in Treating Patients With Recurrent Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0238; NCI-2009-00603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000550975; GOG-0238; GOG-0238 (Other: NRG Oncology); GOG-0238 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Endometrioid Adenocarcinoma, Variant With Squamous Differentiation; Endometrial Mucinous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Recurrent Endometrial Clear Cell Adenocarcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma; Recurrent Endometrial Serous Adenocarcinoma; Recurrent Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Cancer
MeSH Terms: interventions — Radiotherapy, Conformal; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Intensity-Modulated; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (brachytherapy, radiation therapy) (Experimental): Patients undergo EBRT to the pelvis daily on days 1-5 for 5 weeks. After completion of EBRT, patients undergo intracavitary low-dose rate or high-dose rate brachytherapy or low-dose rate interstitial brachytherapy.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Internal Radiation Therapy
- Arm II (brachytherapy, radiation therapy, cisplatin) (Experimental): Patients undergo EBRT as in Arm I and receive cisplatin IV over 1-2 hours on days 1, 8, 15, 22, and 29. Patients then undergo brachytherapy as in Arm I.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Internal Radiation Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm II (brachytherapy, radiation therapy, cisplatin)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Radiation: Internal Radiation Therapy — Given intracavitarily or interstitially
  Other Names: Brachytherapy; Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy; Radiation, Internal

SUMMARY:
This randomized phase II trial studies radiation therapy and cisplatin to see how well they work compared with radiation therapy alone in treating patients with endometrial cancer that has come back. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving radiation therapy together with cisplatin is more effective than radiation therapy alone in treating patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether pelvic radiation therapy with concurrent cisplatin is more promising with respect to progression-free survival than pelvic radiation therapy alone in the treatment of recurrent uterine carcinoma limited to the pelvis and vagina.

SECONDARY OBJECTIVES:

I. To capture the sites of recurrence subsequent to treatment with pelvic radiation with or without concurrent weekly cisplatin in women with recurrent uterine carcinoma.

II. To estimate overall survival of patients with recurrent uterine carcinoma treated with pelvic radiation therapy with or without concurrent weekly cisplatin.

III. To estimate the prognostic significance of the location (central pelvis versus vagina) and size of the recurrence, in addition to the prognostic significance in the salvage setting of the histological subtype, grade, patient age, race, performance status, and the presence of lymph-vascular space involvement of the original tumor at the time of initial hysterectomy.

IV. To evaluate toxicity derived from the combined cisplatin and radiation compared with radiation alone in this patient population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo external-beam radiotherapy (EBRT) to the pelvis daily on days 1-5 for 5 weeks. After completion of EBRT, patients undergo intracavitary low-dose rate or high-dose rate brachytherapy* or low-dose rate interstitial brachytherapy*.

ARM II: Patients undergo EBRT as in Arm I and receive cisplatin intravenously (IV) over 1-2 hours on days 1, 8, 15, 22, and 29. Patients then undergo brachytherapy* as in Arm I.

NOTE: *IMRT boost is allowed for patients who are not candidates for brachytherapy. IMRT may also be used for the entire course of therapy for the treatment of the whole pelvis and/or the boost in patients not undergoing brachytherapy. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every month for 3 months, 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have undergone complete hysterectomy and bilateral salpingo-oophorectomy at the time of original therapy for their uterine carcinoma
* Patients must have a biopsy with histologically confirmed diagnosis of recurrent endometrial cancer confined to the pelvis and/or vagina and no evidence of extrapelvic disease
* Patients must have endometrial carcinoma including endometrioid adenocarcinoma, adenocarcinoma with squamous differentiation, mucinous adenocarcinoma, squamous cell carcinoma, mixed carcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, and serous adenocarcinoma histologies
* Patients must have no evidence of extrapelvic disease; complete workup staging should be performed prior to initiation of therapy to rule-out presence of metastatic disease; this should include: computed tomography (CT) scan of the thorax with IV contrast, as well as a CT of the pelvis and abdomen with IV and oral (PO) contrast performed using multi-detector CT and equal or less than 5 mm slice thickness; if the patient is unable to tolerate contrast, then magnetic resonance imaging (MRI) with IV gadolinium should be performed; a chest x-ray should be done first, and if abnormal, then a CT scan of the chest should be done
* Primary surgical debulking before protocol therapy is permissible; this would include removal of gross symptomatic disease in the pelvis and/or vagina

  * Exenterative surgery is not permissible; patients with complete resection of gross recurrent disease are eligible
* Patients may have received prior hormone therapy and/or systemic chemotherapy; such therapy must have been completed at least 6 months prior to study entry and the patient has clear evidence of disease subsequent to such therapy; patients must not have received neoadjuvant chemotherapy for the present recurrent disease
* Patients must have Gynecologic Oncology Group (GOG) performance status 0, 1, or 2
* Patients must have an estimated survival greater or equal to 3 months
* Absolute neutrophil count (ANC) >= 1,500/mm^3 , equivalent to Common Toxicity Criteria (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 3.0) grade 1
* Platelets >= 100,000/mm^3 (CTCAE v 3.0 grade 0-1)
* Creatinine =< institutional upper limit normal (ULN), CTCAE v 3.0 grade 0; NOTE: if creatinine > ULN, creatinine clearance must be > 50 mL/min
* Bilirubin =< 1.5 x ULN (CTCAE v 3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 x ULN (CTCAE v 3.0 grade 0-1)
* Alkaline phosphatase =< 2.5 x ULN (CTCAE v 3.0 grade 0-1)
* Neuropathy (sensory and motor) =< CTCAE v 3.0 grade 1
* Patients with ureteral obstruction must undergo stent or nephrostomy tube placement prior to study entry
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Patients with evidence of disease outside of the pelvis, including presence of positive periaortic or inguino-femoral nodes
* Patients who have received previous vaginal, pelvic, or abdominal irradiation
* Patients who received chemotherapy directed at the present recurrence
* Patients with septicemia or severe infection
* Patients who have circumstances that will not permit completion of this study or the required follow-up
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have undergone complete surgical resection of the recurrent tumor and have no evidence of residual disease evaluable clinically and by CT or MRI imaging, following resection
* Patients who have a significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, congestive heart failure, or uncontrolled arrhythmias within 6 months of registration
* Patients with history of active collagen vascular disease
* Patients with GOG performance grade of 3 or 4

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-02-25 (Actual); Primary Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Feddock, Principal Investigator — NRG Oncology
Locations (441):
- United States (439):
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Chattanooga Gynecological Oncology, Chattanooga, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (2):
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment onto this study began February 25, 2008. Enrollment of the study ended August 12, 2020 after 165 patients had been enrolled.
Groups:
- Arm I (Brachytherapy, Radiation Therapy): Whole Pelvis Radiation 4500 cGy in 25 fractions to the whole pelvis (180 cGy/fraction) + Interstitial or Intracavitary Brachytherapy or external beam boost
- Arm II (Brachytherapy, Radiation Therapy, Cisplatin): Whole Pelvis Radiation 4500 cGy in 25 Fractions to the whole pelvis (180 cGy/fraction) + Weekly Cisplatin (40mg/m2/wk) + Interstitial or Intracavitary Brachytherapy or external beam boost
Period: Overall Study
Arm/Group | Arm I (Brachytherapy, Radiation Therapy) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin)
Started | 82 | 83
Completed | 74 | 82
Not Completed | 8 | 1
Not completed — Ineligible by Pathology Review | 8 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and Evaluable
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Brachytherapy, Radiation Therapy) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin) | Total
Number analyzed (Participants) | 74 | 82 | 156
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 16 | 19 | 35
  60-80 years | 49 | 59 | 108
  > 80 years | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 82 | 156
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 65 | 74 | 139
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 5 | 1 | 6
  White | 65 | 74 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Tumor Location [Count of Participants; unit: Participants]
  Both pelvis and vagina | 4 | 7 | 11
  Pelvis only | 7 | 4 | 11
  Vagina only | 63 | 71 | 134
Histology [Count of Participants; unit: Participants]
  Endometrioid, grade 1 - usually considered non-aggressive and have the most favorable outcome. | 48 | 42 | 90
  Endometrioid, grade 2 - more likely to spread outside the uterus. Worse outcome than grade 1. | 16 | 22 | 38
  Endometrioid, grade 3 - usually more aggressive with a worse outcome than lower grade tumors. | 2 | 8 | 10
  Endometrioid, grade unknown | 1 | 0 | 1
  Serous | 2 | 4 | 6
  Clear Cell | 1 | 0 | 1
  Mixed Epithelial | 3 | 2 | 5
  Adenocarcinoma, not specified | 1 | 3 | 4
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Progression or Death.
Description: The number of participants with disease progression or death from study entry to progression or death. Participants who experienced progression or death were reported by treatment arm.
Time Frame: Median follow-up for progression-free survival was 62 months with a maximum of 128 months. Patients were followed from study entry until disease progression, death, or date of last contact
Population: Eligible and evaluable participants who experienced progression or died.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Brachytherapy, Radiation Therapy) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin)
Number analyzed (Participants) | 74 | 82
Participants | 27 | 35

2. Secondary Outcome: Number of Participants That Experienced Death on Study
Description: Overall survival is the period from study entry until death or date of last contact. The treatment regimens were compared with regard to overall survival.
Time Frame: Participants were followed from study entry until death or date of last contact. Median follow-up for overall survival was 62 months with a maximum of 128 months.
Population: Eligible and evaluable participants who died while being followed by study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Brachytherapy, Radiation Therapy) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin)
Number analyzed (Participants) | 74 | 82
Participants | 18 | 21

3. Secondary Outcome: Number of Participants in Select Prognostic Groups Who Experienced Progression or Death on Study.
Description: Participants were put in prognostic groups including baseline factors of tumor location (vagina only vs. all others) and histology (serious and clear cell vs. all others). They were assessed for prognostic associations with progression-free survival. Participant factors were collected at baseline. Participants were followed from study entry until disease progression, death, or date of last contact for progression-free survival.
Time Frame: Median follow-up for progression-free survival was 62 months with a maximum of 128 months.
Population: Eligible and evaluable participants who experienced progression or died.
Measure: Count of Participants; unit: Participants
Groups:
- Prognostic Group 1: Participants with vaginal only and serous or clear cell histology
- Prognostic Group 2: Participants with vaginal only and other histology
- Prognostic Group 3: Participants with other tumor location and serous or clear cell histology
- Prognostic Group 4: Patients with other tumor location and other histology
Arm/Group | Prognostic Group 1 | Prognostic Group 2 | Prognostic Group 3 | Prognostic Group 4
Number analyzed (Participants) | 127 | 7 | 0 | 22
Participants | 45 | 4 | 0 | 13

4. Secondary Outcome: Number of Participants That Experienced Adverse Effects Grade 3 or Higher
Description: Number of treated participants with adverse events of grade 3 or higher. Graded by Common Terminology Criteria for Adverse Events version 3.0. Treated patients were evaluated for adverse events during the treatment period, every month for the first three months after completion of therapy up to 2 years, and then every six months for the next 3 years.
Time Frame: Maximum follow-up for adverse events was 61 months.
Population: Number of participants with reported adverse events of grade 3 or higher.
Measure: Count of Participants; unit: Participants
Groups:
- Treated Regimen I: Treated and eligible patients who received regimen I
- Treated Regimen II: Treated and eligible patients who received Regimen II
Arm/Group | Treated Regimen I | Treated Regimen II
Number analyzed (Participants) | 74 | 76
Participants | 37 | 49

ADVERSE EVENTS:
Time Frame: Treated patients were evaluated for adverse events during the treatment period, every month for the first three months after completion of therapy up to 2 years, and then every six months for the next 3 years. Maximum follow-up for adverse events was 61 months. Deaths were reported up to 5 years after study treatment discontinuation. Median follow up for overall survival was 62 months with a maximum of 128 months.
Arm/Group | Arm I (Brachytherapy, Radiation Therapy) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin)
All-Cause Mortality (participants affected / at risk) | 18/74 | 21/82
Serious Adverse Events (participants affected / at risk) | 3/74 | 12/82
Other Adverse Events (participants affected / at risk) | 72/74 | 76/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Brachytherapy, Radiation Therapy) (N=74) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin) (N=82)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 1
Conduction Abnml: Asystole (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Hemorrhage, Gi - Esophagus (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 0 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Brachytherapy, Radiation Therapy) (N=74) | Arm II (Brachytherapy, Radiation Therapy, Cisplatin) (N=82)
Allergy/Immunology - Other (Immune system disorders) | 0 | 1
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 11
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 1 | 3
Neutrophils (Blood and lymphatic system disorders) | 6 | 37
Platelets (Blood and lymphatic system disorders) | 22 | 47
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 7 | 4
Leukocytes (Blood and lymphatic system disorders) | 34 | 61
Lymphopenia (Blood and lymphatic system disorders) | 11 | 12
Hemoglobin (Blood and lymphatic system disorders) | 27 | 50
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 1 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 3 | 0
Edema: Limb (Blood and lymphatic system disorders) | 15 | 19
Edema: Head And Neck (Blood and lymphatic system disorders) | 0 | 2
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 3
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 1 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 | 0
Pulmonary Hypertension (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 21 | 17
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 1
Cardiac General - Other (Cardiac disorders) | 0 | 1
Cardiac Troponin I (Ctni) (Cardiac disorders) | 1 | 1
Hypotension (Cardiac disorders) | 1 | 2
Inr (Vascular disorders) | 0 | 1
Coagulopathy - Other (Vascular disorders) | 0 | 1
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 3 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 15 | 12
Hemorrhage, Gi - Rectum (Vascular disorders) | 9 | 9
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 2 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1 | 1
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Anus (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 1 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 2
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 4
Phlebitis (Vascular disorders) | 0 | 1
Constitutional Symptoms - Other (General disorders) | 4 | 2
Sweating (General disorders) | 1 | 2
Weight Gain (General disorders) | 2 | 1
Patient Odor (General disorders) | 0 | 1
Fever (General disorders) | 1 | 5
Weight Loss (General disorders) | 11 | 6
Obesity (General disorders) | 0 | 1
Rigors/Chills (General disorders) | 2 | 4
Fatigue (General disorders) | 52 | 64
Insomnia (General disorders) | 10 | 18
Pain - Other (General disorders) | 7 | 11
Pain: Urethra (General disorders) | 9 | 8
Pain: Perineum (General disorders) | 2 | 0
Pain: Pelvis (General disorders) | 12 | 6
Pain: Breast (General disorders) | 1 | 0
Pain: Vagina (General disorders) | 10 | 5
Pain: Chest /Thorax Nos (General disorders) | 0 | 1
Pain: Chest Wall (General disorders) | 0 | 4
Pain: Head/Headache (General disorders) | 6 | 18
Pain: Neck (General disorders) | 0 | 2
Pain: Intestine (General disorders) | 1 | 0
Pain: Extremity-Limb (General disorders) | 6 | 7
Pain: Buttock (General disorders) | 3 | 1
Pain: Back (General disorders) | 12 | 16
Pain: Joint (General disorders) | 11 | 12
Pain: Bone (General disorders) | 1 | 1
Pain: Lymph Node (General disorders) | 0 | 1
Pain: Bladder (General disorders) | 2 | 1
Pain: Pain Nos (General disorders) | 5 | 6
Pain: Stomach (General disorders) | 0 | 2
Pain: Rectum (General disorders) | 6 | 4
Pain: Abdominal Pain Nos (General disorders) | 26 | 14
Pain: Skin (General disorders) | 1 | 0
Pain: Lip (General disorders) | 1 | 0
Pain: Middle Ear (General disorders) | 1 | 1
Pain: External Ear (General disorders) | 0 | 2
Pain: Cardiac/ Heart (General disorders) | 0 | 1
Pain: Muscle (General disorders) | 1 | 1
Pain: Anus (General disorders) | 1 | 2
Pain: Neuralgia (General disorders) | 1 | 1
Flu-Like Syndrome (General disorders) | 0 | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 0 | 2
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 5 | 5
Dermatitis - Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Bruising (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 2
Atrophy, Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis - Radiation (Skin and subcutaneous tissue disorders) | 11 | 7
Telangiectasia (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Burn (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 3
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 2 | 0
Hot Flashes (Endocrine disorders) | 3 | 5
Diabetes (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1
Enteritis (Gastrointestinal disorders) | 1 | 2
Proctitis (Gastrointestinal disorders) | 6 | 6
Flatulence (Gastrointestinal disorders) | 1 | 6
Fistula, Gi - Rectum (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 9 | 7
Ulcer,gi - Rectum (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 5
Ileus (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Distention (Gastrointestinal disorders) | 4 | 5
Taste Alteration (Gastrointestinal disorders) | 5 | 15
Incontinence, Anal (Gastrointestinal disorders) | 2 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 0 | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2 | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 3 | 2
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 0 | 6
Vomiting (Gastrointestinal disorders) | 10 | 18
Anorexia (Gastrointestinal disorders) | 19 | 24
Dehydration (Gastrointestinal disorders) | 1 | 10
Constipation (Gastrointestinal disorders) | 21 | 29
Nausea (Gastrointestinal disorders) | 28 | 53
Gastrointestinal - Other (Gastrointestinal disorders) | 5 | 6
Diarrhea (Gastrointestinal disorders) | 62 | 65
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 0 | 2
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 5 | 4
Inf Unknown Anc: Blood (Infections and infestations) | 1 | 1
Infection - Other (Infections and infestations) | 3 | 5
Inf Unknown Anc: Vagina (Infections and infestations) | 1 | 1
Inf Unknown Anc: Eye Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 6 | 5
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1 | 1
Inf Unknown Anc: Dental-Tooth (Infections and infestations) | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 0
Ast (Metabolism and nutrition disorders) | 5 | 8
Gfr (Metabolism and nutrition disorders) | 1 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 3 | 4
Cholesterol,serum High (Metabolism and nutrition disorders) | 1 | 2
Proteinuria (Metabolism and nutrition disorders) | 3 | 2
Creatinine (Metabolism and nutrition disorders) | 9 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 14
Ggt (Metabolism and nutrition disorders) | 0 | 1
Alt (Metabolism and nutrition disorders) | 10 | 11
Alkaline Phosphatase (Metabolism and nutrition disorders) | 4 | 3
Bilirubin (Metabolism and nutrition disorders) | 1 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 8
Hyponatremia (Metabolism and nutrition disorders) | 4 | 21
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 11 | 23
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 26
Hypokalemia (Metabolism and nutrition disorders) | 14 | 19
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 29
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 6 | 3
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 6 | 9
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Psychosis (Nervous system disorders) | 0 | 1
Neurology - Other (Nervous system disorders) | 2 | 1
Apnea (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Mood Alteration - Euphoria (Nervous system disorders) | 1 | 0
Mood Alteration - Depression (Nervous system disorders) | 10 | 7
Mood Alteration - Anxiety (Nervous system disorders) | 8 | 11
Mood Alteration - Agitation (Nervous system disorders) | 4 | 3
Tremor (Nervous system disorders) | 0 | 1
Speech Impairment (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 6 | 0
Dizziness (Nervous system disorders) | 6 | 10
Neuropathy-Sensory (Nervous system disorders) | 10 | 18
Neuropathy-Motor (Nervous system disorders) | 0 | 2
Ocular/Visual - Other (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 0
Blurred Vision (Eye disorders) | 3 | 6
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Renal/Genitourinary - Other (Renal and urinary disorders) | 10 | 8
Stricture, Anastomotic, Gu - Vagina (Renal and urinary disorders) | 0 | 2
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Leak, Gu - Urethra (Renal and urinary disorders) | 2 | 0
Cystitis (Renal and urinary disorders) | 5 | 9
Urinary Color Change (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 6
Obstruction, Gu - Urethra (Renal and urinary disorders) | 1 | 0
Incontinence, Urinary (Renal and urinary disorders) | 8 | 15
Fistula, Gu - Vagina (Renal and urinary disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 5 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 22 | 21
Libido (Reproductive system and breast disorders) | 0 | 1
Irregular Menses (Reproductive system and breast disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 4 | 0
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 6 | 8
Vaginitis (Reproductive system and breast disorders) | 5 | 2
Vaginal Stenosis (Reproductive system and breast disorders) | 6 | 4
Vaginal Mucositis (Reproductive system and breast disorders) | 4 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 17 | 14
Intra-Op Injury: Bone (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT00492778/Prot_SAP_000.pdf